CLINICAL TRIAL: NCT07358702
Title: Comparison of Body Awareness, Respiratory Muscle Strength, Kinesiophobia, Central Sensitization, Functional Status and Sleep Quality in Sedentary and Non-Sedentary Fibromyalgia Individuals
Brief Title: Sedentary Status and Multidimensional Outcomes in Fibromyalgia
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Izmir Democracy University (Other)
Responsible Party: Principal Investigator, Betül Taşpınar, Prof.Dr., Izmir Democracy University
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: Sedentary FMS-35
Record Dates: First submitted 2026-01-13; First posted 2026-01-22 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Fibromyalgia; Sedentary Behavior; Kinesiophobia; Central Sensitisation
Keywords: Fibromyalgia Syndrome; Sedentary Behavior; Functional Status
MeSH Terms: conditions — Fibromyalgia; Sedentary Behavior; Kinesiophobia

STUDY DESIGN:
Intervention Model Description: Individuals diagnosed with fibromyalgia syndrome will be categorized into two groups based on their physical activity level: sedentary and non-sedentary. The groups will be compared in terms of body awareness, respiratory muscle strength, kinesiophobia, central sensitization, functional status, and sleep quality. The aim is to evaluate the differences in these multidimensional clinical parameters between sedentary and non-sedentary individuals with fibromyalgia.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sedentary Fibromyalgia Group (Other): Individuals diagnosed with fibromyalgia syndrome who meet the criteria for sedentary behavior.
  Interventions: Other: Assessment Only
- Non-Sedentary Fibromyalgia Group (Other): Individuals diagnosed with fibromyalgia syndrome who do not meet the criteria for sedentary behavior.
  Interventions: Other: Assessment Only

INTERVENTIONS:
Other: Assessment Only — No therapeutic intervention will be applied in this study. Participants will undergo a comprehensive assessment to evaluate clinical and functional characteristics. Assessments will include body awareness, respiratory muscle strength, kinesiophobia, central sensitization, functional status, sleep quality, and physical activity level. All evaluations will be conducted at a single time point using validated clinical measurement tools and self-reported questionnaires. The purpose of these assessments is to compare sedentary and non-sedentary individuals with fibromyalgia syndrome in terms of multidimensional clinical outcomes.

SUMMARY:
Fibromyalgia syndrome (FMS) is a chronic condition characterized by widespread musculoskeletal pain, fatigue, sleep disturbances, and functional limitations. Pain, fatigue, and fear of movement often lead individuals with FMS to adopt sedentary behaviors, which may further exacerbate symptoms and reduce physical capacity. Factors such as impaired body awareness, reduced respiratory muscle strength, kinesiophobia, central sensitization, poor functional status, and sleep disturbances play an important role in disease severity and quality of life in individuals with FMS.

Although physical inactivity is common in fibromyalgia, limited evidence exists regarding the differences in these multidimensional clinical parameters between sedentary and non-sedentary individuals with FMS. Therefore, the aim of this study is to compare body awareness, respiratory muscle strength, kinesiophobia, central sensitization, functional status, and sleep quality between sedentary and non-sedentary individuals diagnosed with fibromyalgia syndrome. The findings of this study may contribute to a better understanding of the impact of sedentary behavior on clinical outcomes in fibromyalgia and help guide more comprehensive and individualized rehabilitation approaches.

DETAILED DESCRIPTION:
Fibromyalgia syndrome (FMS) is a chronic pain condition characterized by widespread musculoskeletal pain, sleep disturbances, and fatigue. Along with other symptoms such as joint stiffness, depression, anxiety, and cognitive dysfunction, FMS restricts daily life, negatively affects physical activity, and reduces individuals' ability to cope with daily demands. Moreover, FMS can lead to reduced productivity, work-related disability, and increased healthcare costs. As a result, patients experience limitations in activities of daily living and overall functional capacity. As a chronic pain condition, FMS may contribute to impaired functional capacity through the adoption of sedentary behaviors. Pain and fatigue associated with FMS often lead to physical inactivity, resulting in muscle deconditioning and, consequently, increased pain and fatigue, creating a vicious cycle. FMS affects approximately 2-6% of the global population and is the second most common rheumatologic disorder after osteoarthritis. However, the pathogenesis of the disease has not yet been fully elucidated.

Body awareness refers to the ability to perceive bodily sensations, movements, and the relationship between the body and its environment. In individuals with FMS, body awareness is often impaired, leading to difficulties in recognizing and interpreting bodily signals related to pain, fatigue, and stress. This impairment in body awareness may exacerbate symptoms and hinder the implementation of effective coping strategies. Enhanced body awareness allows patients to identify factors that trigger pain and to develop more effective coping mechanisms. Previous studies have demonstrated that therapeutic approaches focusing on body awareness are beneficial in reducing pain levels and improving movement quality in individuals with FMS.

Body awareness is also associated with psychological factors commonly observed in individuals with FMS, such as anxiety and depression. It has been reported that as body awareness increases, individuals with FMS are better able to analyze their emotional responses to their physical condition, which may help reduce anxiety levels. Furthermore, studies have shown that interventions aimed at improving body awareness result in positive changes in psychological functioning, including reductions in anxiety and depression, in individuals with FMS.

Compared with healthy individuals, people with FMS exhibit lower respiratory muscle strength and endurance. Studies in the literature indicate that maximal inspiratory pressure and maximal expiratory pressure-important indicators of respiratory muscle performance-are reduced in individuals with FMS. This reduction can cause difficulty in breathing during physical activities, contributing to a persistent cycle of fatigue and weakness. A correlation has been observed between respiratory muscle strength and the severity of FMS symptoms. Previous studies have demonstrated that reduced inspiratory muscle strength is associated with a higher number of tender points, greater fatigue severity, and decreased thoracic mobility.

Participation in physical activities among individuals with FMS is often limited due to pain and fatigue, and the resulting increase in physical inactivity further reduces respiratory muscle strength. Interventions aimed at improving respiratory muscle strength have been shown to enhance exercise tolerance, physical function, and quality of life, while also reducing pain and fatigue.

Kinesiophobia, defined as an excessive and debilitating fear of movement or physical activity, plays a significant role in disease management and the development of coping strategies in individuals with FMS. Kinesiophobia is observed in more than 38% of individuals with FMS. High levels of kinesiophobia have been associated with increased pain intensity, disease activity, and depression severity, as well as decreased physical activity and quality of life. Individuals with FMS often perceive pain as a threat, leading to increased avoidance of physical activity. As a result, fear-avoidance behaviors develop, which exacerbate FMS symptoms and increase levels of disability.

Central sensitization refers to increased responsiveness of the central nervous system (CNS) to stimulation. This phenomenon occurs when the CNS becomes excessively sensitive to sensory input, resulting in heightened pain perception in response to normally non-painful stimuli (allodynia) or exaggerated responses to painful stimuli (hyperalgesia). Although central sensitization is not specific to FMS, it plays a crucial role in its pathophysiology. Central sensitization involves complex neurobiological processes, including alterations in neurotransmitter levels, neuronal pathways, and brain structure and function. These changes are influenced by genetic predisposition, previous injuries, stress, and psychological factors.

Fibromyalgia is generally considered a central sensitization syndrome. Chronic pain in individuals with FMS is believed to arise primarily from central sensitization rather than peripheral tissue injury or inflammation. Proinflammatory cytokines are frequently elevated in patients with fibromyalgia and contribute to the development of central sensitization. These cytokines may activate glial cells in the CNS, leading to persistent pain perception.

Sleep disturbances are a common symptom in individuals with FMS. Patients frequently report difficulty falling asleep, frequent nighttime awakenings, and waking up feeling unrefreshed. These disturbances are often attributed to alterations in normal brain wave activity, which prevent the transition into deep sleep stages necessary for physical restoration and mental clarity. Individuals with FMS may also report a subjective sensation of swelling in muscles and joints, although this finding is not typically observed during physical examination.

Approximately 90% of individuals with FMS experience sleep disorders, including insomnia, restless legs syndrome, and sleep apnea. A bidirectional relationship exists between sleep and pain in FMS. Poor sleep quality increases pain sensitivity and lowers pain thresholds, while increased pain severity exacerbates sleep disturbances, creating a vicious cycle. In addition to its effects on pain severity, poor sleep quality has been shown to negatively impact cognitive function, fatigue, anxiety, and depression.

Physical activity is defined as any bodily movement produced by skeletal muscles that results in energy expenditure and includes both activities of daily living and planned exercise. Studies have shown that individuals with FMS have lower levels of physical activity compared with healthy individuals. Only 37% of individuals with FMS meet the guideline-recommended level of at least 150 minutes of moderate-to-vigorous physical activity per week. Additionally, individuals with FMS take an average of 5,663.7 steps per day, which is below the recommended daily target of 6,000 steps. Compared with healthy individuals, they also spend less time engaging in daily activities such as leisure and transportation. Approximately 36.6% of individuals with fibromyalgia are classified as inactive, while an additional 45.1% are considered insufficiently active.

The primary barriers to physical activity in individuals with FMS include persistent fatigue, pain, fear of symptom exacerbation with exertion, disability, mood disorders, low self-efficacy for movement, and inadequate social support. Chronic pain and fatigue lead individuals with FMS to avoid physical activity. Many individuals believe that physical activity will worsen their symptoms, resulting in fear-avoidance behaviors. The combination of inactivity and pain often leads to reduced muscle strength, making activities of daily living more difficult. Studies have demonstrated that individuals with FMS exhibit decreased physical conditioning, low cardiorespiratory endurance, and reduced muscle strength and endurance. Despite these barriers, regular physical activity provides numerous benefits for individuals with FMS.

Physical activity has been reported to alleviate FMS symptoms by increasing the release of neurotransmitters such as endorphins and serotonin. Additionally, physical activity plays an important role in influencing fatigue both directly and indirectly through regulation of the hypothalamic-pituitary-adrenal axis and autonomic nervous system function. When physical activity is performed in group settings, social interaction may enhance well-being and reduce psychological distress, thereby improving quality of life. It has been demonstrated that engaging in light- to moderate-intensity physical activity and exercise two to three times per week increases muscle strength, reduces pain, improves flexibility, and enhances quality of life in individuals with FMS.

Although studies have compared physical activity levels between individuals with FMS and healthy controls, there is currently no study comparing body awareness, respiratory muscle strength, kinesiophobia, central sensitization, functional status, and sleep quality between sedentary and non-sedentary individuals with fibromyalgia.

ELIGIBILITY:
Inclusion Criteria - Sedentary Fibromyalgia Participants

* Physical activity level below 600 MET-min/week according to the International Physical Activity Questionnaire (IPAQ)
* Diagnosis of fibromyalgia according to the 2016 ACR criteria
* Age between 18 and 65 years
* Ability to understand and respond to study assessments

Exclusion Criteria - Sedentary Fibromyalgia Participants

* Conditions posing risk during assessments, including unstable angina, decompensated heart failure, or myocardial infarction within the past month
* Uncontrolled diabetes, hypertension >180/110 mmHg, and/or severe neuropathy
* Diagnosed severe cognitive impairment
* Pregnancy or suspected pregnancy Inclusion Criteria - Non-Sedentary Fibromyalgia Participants
* Physical activity level above 600 MET-min/week according to the IPAQ
* Diagnosis of fibromyalgia according to the 2016 ACR criteria
* Age between 18 and 65 years
* Ability to understand and respond to study assessments

Exclusion Criteria - Non-Sedentary Fibromyalgia Participants

* Conditions posing risk during assessments, including unstable angina, decompensated heart failure, or myocardial infarction within the past month
* Uncontrolled diabetes, hypertension >180/110 mmHg, and/or severe neuropathy
* Diagnosed severe cognitive impairment
* Pregnancy or suspected pregnancy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2026-05-15 (Estimated); Primary Completion 2026-10-15 (Estimated); Study Completion 2027-01-15 (Estimated)

PRIMARY OUTCOMES:
International Physical Activity Questionnaire (IPAQ) - Short Form | Baseline
  The International Physical Activity Questionnaire (IPAQ) is commonly used to assess physical activity. In this study, the 7-item short form of the IPAQ will be used. The questionnaire evaluates the number of days and duration over the past 7 days in which participants performed vigorous physical activity, moderate physical activity, and walking for at least 10 minutes per session. Total physical activity is calculated by multiplying the duration and frequency of each activity by its MET value: 8 MET for vigorous, 4 MET for moderate, and 3.3 MET for walking. Sedentary time is not included in the calculation. The weekly MET score is summed across all activities: <600 MET-min/week is considered inactive, 601-3,000 MET-min/week moderately active, and >3,000 MET-min/week active
Mindful Attention Awareness Scale (MAAS) | Baseline
  The MAAS is a 15-item scale measuring the general tendency to be aware of and attentive to present-moment experiences. The scale is unidimensional, yielding a single total score, where higher scores indicate greater mindfulness. Items are rated on a 6-point Likert scale from 1 (almost always) to 6 (almost never).
Postural Awareness Scale (PAS) | Baseline
  The Postural Awareness Scale evaluates individuals' postural awareness and efforts to regulate their posture. It consists of two factors and a total of 11 items. Total scores range from 11 to 77, with higher scores indicating better postural awareness.
Fibromyalgia Impact Questionnaire (FIQ) | Baseline
  The Fibromyalgia Impact Questionnaire (FIQ) assesses functional status in fibromyalgia patients. The FIQ evaluates 10 domains: physical function, feeling well, work difficulty, work missed, pain, fatigue, morning tiredness, stiffness, anxiety, and depression. Excluding the "feeling well" domain, lower scores indicate better function. The questionnaire is patient-reported and takes approximately 5 minutes to complete, with a total score of 100. Physical Function Subscale: 11 questions scored 0-3, summed and averaged, then multiplied by 3.33 (range 0-33).Feeling Well Subscale: Reverse-scored, average multiplied by 1.43 (range 0-7).Work Missed Subscale: Directly scored, multiplied by 1.43. Other domains: Scored 0-10 per item; higher scores indicate greater impairment. All scores are summed to obtain a total FIQ score.
Tampa Scale of Kinesiophobia (TSK) | Baseline
  The Tampa Scale for Kinesiophobia (TSK) was originally developed to assess fear of movement. The scale has 17 items, rated on a 4-point Likert scale (1 = strongly disagree to 4 = strongly agree). Items 4, 8, 12, and 16 are reverse-scored. Higher total scores indicate higher kinesiophobia.
Central Sensitization Inventory (CSI) | Baseline
  The CSI assesses symptoms related to central sensitization in individuals with chronic pain. It consists of two parts: Part A evaluates 25 somatic and psychosocial symptoms commonly associated with central sensitization; Part B identifies medical conditions known to be related to central sensitization (not scored). Total scores are out of 100, with ≥40 indicating the presence of central sensitization.
Pittsburgh Sleep Quality Index (PSQI) | Baseline
  The PSQI is a 24-item self-report questionnaire evaluating sleep quality and disturbances. The first 19 items are self-rated, and the remaining 5 are answered by a partner or roommate but are not included in scoring. Higher total scores indicate worse sleep quality. Seven subcomponents are scored 0-3: subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleep medication, and daytime dysfunction. Total scores range from 0-21; scores ≥5 indicate poor sleep quality
Respiratory Muscle Strength Assessment | Baseline
  Respiratory muscle strength will be measured using the Cosmed Pony FX spirometer. Maximal inspiratory pressure (MIP) and maximal expiratory pressure (MEP) will be assessed. MIP: Participant performs maximal expiration in a seated position, followed by maximal inspiration against a closed airway for 1-3 seconds. MEP: Participant performs maximal inspiration, followed by maximal expiration against a closed airway for 1-3 seconds. Three measurements will be taken, and the best value will be recorded. Age- and sex-specific reference values will be used.

CONTACTS AND LOCATIONS:
Overall Officials: Onur Engin, Asst.Prof., Principal Investigator — Izmir Democracy University; Ayşe Sezgi Kızılırmak Karataş, Asst.Prof, Principal Investigator — Izmir Democracy University; Büşra Aydın, std., Principal Investigator — Izmir Democracy University; Öykü Dündar, std., Principal Investigator — Izmir Democracy University; Turna Sümen, std., Principal Investigator — Izmir Democracy University; Nalan Anık, std., Principal Investigator — Izmir Democracy University; Kader İliman, std., Principal Investigator — Izmir Democracy University; Fadıma Kılıç, std., Principal Investigator — Izmir Democracy University
Locations (1):
- Betül TAŞPINAR, Konak, İ̇zmi̇r, Turkey (Türkiye)